CLINICAL TRIAL: NCT00965198
Title: Comparison of a Novel Silver-Coated Catheter Access Device and a Standard Catheter Access Device: A Dual Center Cross-Over Study
Brief Title: Comparison of Infection Rates Among Patients Using Two Catheter Access Devices
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Jesse Thomas Jacob, Investigator, Emory University
Other Study IDs: IRB00016682; B16682 (Other: Other)
Record Dates: First submitted 2009-07-16; First posted 2009-08-25 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Catheter-Related Infections; Bacteremia
Keywords: Catheters, Indwelling; Biofilms
MeSH Terms: conditions — Catheter-Related Infections; Bacteremia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples for biofilm analysis may be banked for further study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Clearlink Arm, EUH: Standard catheter access device at Emory University Hospital
- VLINK Arm, EUHM: Novel, silver-coated catheter access device at Emory University Hospital Midtown
- Clearlink, EUM: Standard catheter access device at at Emory University Hospital Midtown
- VLINK Arm, EUH: Novel, silver-coated catheter access device at Emory University Hospital

SUMMARY:
Intravenous catheters are placed in nearly every hospitalized patient. These catheters, since they are breaks in skin integrity, are potential sources of infection that occur in the bloodstream. Bloodstream infections can result in higher rates of death and lengths of hospital stay, as well as increase healthcare costs. Blood is drawn or medications delivered through a catheter access device attached to the catheter. In looking at new ways to decrease infections associated with healthcare, the investigators plan to test whether the use of a silver-coated catheter access device (VLINK) compared to the standard, non-coated device (CLEARLINK) can reduce infection rates. These devices are identical in design other than the silver coating of the VLINK, that imparts a brown color to the device. Silver can prevent the growth of bacteria inside the device (biofilm formation) in the laboratory, but this has never been proven in patients.

The investigators propose to do a crossover study in two Emory-owned hospitals (Emory University Hospital and Emory University Hospital at Midtown), anticipated to last 10 months. Currently, both types of devices, (standard and silver-coated) are FDA approved for clinical use and are in use at both hospitals. The investigators plan to have each hospital use only one type of catheter access device for a period of time (approximately 5 months), and then switch ("crossover") to other type of device for the rest of the study. All patients admitted to either hospital (excluding newborns and patients with infections attributed to hemodialysis catheters) will be enrolled since both devices meet the standard of care. During the study, the infection prevention department, as a continuing part of their regular duties will measure infection rates. A small subset of catheters that are removed during routine clinical care (none will be taken out solely for the study) will be sent to CDC to determine the amount of bacteria inside catheters and catheter access devices (look for biofilm). Finally, the microbiology lab, again as part of its routine function will determine the rate at which blood cultures are falsely positive. All of these measures will be compared using statistical methods to see if there is a difference between the standard and silver-coated catheter access devices.

In undertaking this study, the investigators will be using a type of vascular access device (valve, not positive pressure) already in use in both hospitals and not changing the delivery of care to patients while, in a rigorous, systematic manner, obtaining samples and data for analysis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the two participating hospitals.

Exclusion Criteria:

* Catheter-associated infections attributed to hemodialysis catheters.
* Neonates and children.
* Known silver allergy or hypersensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nearly all hospitalized patients require some form of indwelling IV catheter as part of routine care, and approximately 20% of patient-days include central lines. All adult patients admitted to 2 Emory affiliated hospitals (Emory University Hospital and Emory University Hospital Midtown) during the study period will be included in the study population.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
central-line associated bloodstream infections rate per 1,000 central line-days | 1 year

SECONDARY OUTCOMES:
intravenous catheter related bloodstream infection rate per 1,000 patient-days | 1 year
colony counts per device analyzed (biofilm analysis) | devices due to be changed at day 7
false positive blood culture rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James P Steinberg, MD, Principal Investigator — Emory University; Jesse T Jacob, MD, Study Director — Emory University; Sheri Chernetsky Tejedor, MD, Study Director — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia